CLINICAL TRIAL: NCT02415829
Title: Efficacy and Safety of Oxaliplatin Combined With Capecitabine as Neoadjuvant Chemotherapy for Locally Advanced Colon Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ye Xu, professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1501143-1
Record Dates: First submitted 2015-03-30; First posted 2015-04-14 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Colorectal Cancer
Keywords: Neoajuvant chemotherapy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Capecitabine; Oxaliplatin

ARMS (1):
- Neoadjuvant chemotherapy (Experimental): A total of 55 cases of locally advanced colon cancer will be enrolled in this arm. After radiological staging, patients were treated first with 3 cycles of neoadjuvant chemotherapy consisting of oxaliplatin, 130 mg/m² on day 1, with capecitabine, 1000 mg/m² twice daily for 14 days every 3 weeks (the XELOX regimen), followed by tumor resection, and then with another 5 cycles of adjuvant chemotherapy with the XELOX regimen. Radiological response was evaluated after 2 cycles of neoadjuvant chemotherapy . A total of 3 cycles neoadjuvant chemotherapy was completed unless there was unacceptable toxicity, emergency operation condition or tumor progression during the period. Tumor responses, toxicities, and surgical complications were recorded. The pathological tumor response in the primary tumor was evaluated according to tumor regression grade (TRG) score.
  Interventions: Drug: capecitabine plus oxaliplatin

INTERVENTIONS:
Drug: capecitabine plus oxaliplatin — The neoadjuvant chemotherapy consisted of oxaliplatin, 130 mg/m² on day 1, with capecitabine, 1000 mg/m² twice daily for 14 days every 3 weeks (the XELOX regimen)

SUMMARY:
The study aims to identify the efficacy and safety of capecitabine plus oxaliplatin (XELOX) in patients with local advanced colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Performance status (ECOG) 0~2
2. Histologically confirmed colon cancer.
3. No prior treatment
4. CT-defined T4 or lymph node-positive colon cancer
5. Neutrophils ≥ 1.5 x 109/L, platelets ≥ 100 x 109/L, and hemoglobin ≥ 8 g/dL Bilirubin level ≤ 1.0 x ULN
6. AST and ALT < 1.5 x ULN
7. Serum creatinine ≤ 1.0 x ULN
8. Life expectancy of ≥ 3 months
9. Signed written informed consent

Exclusion Criteria:

1. Final stage with cancer cachexia
2. Allergy for capecitabine or oxaliplatin
3. Any evidence of extrahepatic metastases and/or primary tumor recurrence
4. Severe organ failures or diseases, including: clinically relevant coronary disease, cardiovascular disorder or myocardial infarction within 12 months before study entry, severe psychiatric illness, severe infection and DIC

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2014-11; Primary Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
The tumor regression grade of all the patients enrolled | from the first cycle of treatment (day one) to tumor resection

SECONDARY OUTCOMES:
Number of Participants receiving complete tumor resection | From date of randomization until the date of the last patients receiving the surgery
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | from the first cycle of treatment (day one) to six month after the last cycle

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Colorectal Surgery Fudan University Shanghai Caner Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Liu F, Yang L, Wu Y, Li C, Zhao J, Keranmu A, Zheng H, Huang D, Wang L, Tong T, Xu J, Zhu J, Cai S, Xu Y. CapOX as neoadjuvant chemotherapy for locally advanced operable colon cancer patients: a prospective single-arm phase II trial. Chin J Cancer Res. 2016 Dec;28(6):589-597. doi: 10.21147/j.issn.1000-9604.2016.06.05. PMID 28174487